CLINICAL TRIAL: NCT07336056
Title: Safety Profile of High-Frequency Use of a Remote Electrical Neuromodulation (REN) Wearable Device for Migraine Treatment
Brief Title: Nerivio Efficacy Under High-Frequency Use
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RWE-013
Record Dates: First submitted 2026-01-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: treatment of migraine; Remote Electrical Neuromodulation; Nerivio
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: REN treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nerivio users who treated with nerivio in patterns acceding the indication for use (Active Comparator): Nerivio users who treatedfrequantly with Nerivio under the following regiemes:
  1. - Multiple treatments per day: defined as administrating 4 or more full treatments on a single day.
  2. - Administrating at least one full treatment on 25 or more days within a 28-day period. For each patient, all possible 28-day windows containing at least 25 treatment days were identified.
  Interventions: Device: Nerivio (REN device)

INTERVENTIONS:
Device: Nerivio (REN device) — Remote electrical neuromodulation (REN) device for the acute treatment of migraines. The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application

SUMMARY:
This is a Post-marketing study investigating the impact of frequant usage with Nerivio on the safety profile of Remote Electrical Neuromodulation (REN) for the treatment of migraine.

This study assessed the safety and tolerability of REN when used at frequencies exceeding the labeled indication.

DETAILED DESCRIPTION:
The REN device (Nerivio by Theranica, ISRAEL) is a neuromodulation device approved by the FDA for acute and/or preventive treatment of migraine in patients 8 years old and above. It is a wearable device applied to the upper arm. It stimulates C and Aδ noxious fibers using a modulated, symmetrical, biphasic, square pulse with a pulse width of 400 μs and up to 40 mA output current, which the patient can adjust. The REN device is operated by a designated app that is downloaded to the user's phone prior to first use of the Nerivio device. As part of the sign-up process for the Nerivio app, all patients accept the terms of use, which specify that providing personal information is done on their own free will and that their de-identified data may be used for research purposes. Users are not obligated to provide personal information and could treat without providing any feedback.

The app includes a secure, personal migraine diary, which enables patients to record and track their migraines and other headaches. At the beginning of each treatment, and again at 2 hours after the start of treatment, patients are prompted to record their symptoms, including pain level (none, mild, moderate, severe), functional disability (None, Mild limitation, Moderate limitation, Severe limitation), and an indication of which medications, if any, were taken within that 2-hour time window.

Post-marketing surveillance is designed to assess the safety, utilization, and efficacy in larger and more diverse populations and in various real-world environments and situations. As a digital therapeutic device (i.e., electroceutical), the REN device enables prospective collection of electronic patient-reported outcomes in real-world clinical practice.

According to the indication, acute treatment with REN should start as early as possible once a migraine attack begins, or every other day for preventive treatment. Given that the instruction is to use "as needed", empowering patients to find the best treatment regime that works for them, real-world treatment patterns may deviate from the approved indication. As patients are not limited in the number of treatments they can conduct per day, nor by the number of treatment days per month, some patients who experience frequent and severe headaches and associated-symptoms, have adopted more frequent treatment regimens, including multiple treatments within a single day, daily use, or a combination of both patterns. The safety profile of REN under such frequent use conditions has not been systematically evaluated.

The objective of this study is to assess the safety and tolerability of the REN wearable device when used at frequencies exceeding the labeled indication, defined as either multiple treatments per day or daily use, using real-world data from patients who were prescribed the device as part of their routine migraine care.

ELIGIBILITY:
Inclusion Criteria:

* Nerivio user
* Treated at least 4 times in a singe day, Or: treated at leastonce in 25 out of 28 consecutive days

ExclusiveCriteria:

* None

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of Nerivio treatment | up to 5 years
  Rate of serious adverse events, adverse events and device-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alit Stark-Inbar, PhD, Principal Investigator — Theranica
Locations (1):
- Theranica USA Inc, Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No